CLINICAL TRIAL: NCT04433117
Title: Bone Quality and Quantity in the Maxillary Sinus Grafted With Xenograft or Synthetic Bone Substitute: A Radiographic and Histomorphometric Randomized Controlled Clinical Study
Brief Title: Bone Material Comparison in Maxillary Sinus Augmentation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohanad Al-Sabbagh (Other)
Responsible Party: Sponsor-Investigator, Mohanad Al-Sabbagh, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 58349
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Bone Resorption; Sequela; Tooth Extrusion
Keywords: Sinus pneumatization; Socket preservation; Sinus augmentation
MeSH Terms: interventions — Bio-Oss

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial. Entails 2 groups of subjects which will be randomly assigned. Group 1 will be the control group, and group 2 is test group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Other): Control group in this study will comprise of 10 subjects and will receive Bio-Oss xenograft bone material.
  Interventions: Biological: Bio-Oss
- Test Group (Experimental): The test group in this study will comprise of 10 subjects and will receive Shefabone synthetic bone substitute.
  Interventions: Biological: Shefabone

INTERVENTIONS:
Biological: Shefabone — Silica-calcium phosphate composite.
  Arms: Test Group
Biological: Bio-Oss — Xenograft Bone substitute. Bone from animals.
  Other Names: Bio-Oss by Geistlich
  Arms: Control Group

SUMMARY:
Hard and soft tissue deficiencies of an alveolar ridge arise as sequelae of tooth extraction when socket preservation is not applied. In addition, extraction of posterior maxillary teeth causes pneumatization of the maxillary sinus in relation to other fixed landmarks such as the teeth. These anatomic sinus limitations and alveolar bone deficiencies are the main challenges for dental implant placement. Different bone substitutes have been used to augment bone in pneumatized maxillary sinuses.

Scaffolding materials such as xenografts or synthetics substitutes have been proven to be a viable alternative.

Xenografts are obtained from nonhuman species and serve as a scaffold for the formation of new bone (osteoconduction). Histologic evaluation of maxillary sinuses grafted with xenografts revealed newly formed bone to be mostly woven bone with some remodeling to lamellar bone. These histologic findings reaffirm the osteoconductive ability of xenografts when used as the sole grafting material in maxillary sinus augmentation. Xenografts appear to be an effective method for maxillary sinus grafting and demonstrate limited resorption over time. Sinuses augmented with synthetic bone substitute (SBS) also appear to successfully integrate based on recent histomorphometric studies. Vascularization and trabecular bone formation in sinuses grafted with SBS has been previously demonstrated. One type of SBS includes porous granules of bioactive and resorbable silica-calcium phosphate nanocomposite (ShefaBone). ShefaBone grafts offer a novel alternative that can potentially unite the 3 salient bone-forming properties (osteoinduction, osteoconduction, and osteogenesis). ShefaBone has unique properties including: 1) bioactivity 2) bioresorbablility, and 3) allowing for the uptake of calcium ions from the physiological solution and releasing phosphate and silicate ions which aid in bone formation. A material with such properties will substitute bone in a more controlled and effective combination that can be obtained in many clinical situations, without the disadvantages found with autograft. ShefaBone has demonstrated successful regenerative properties for bony defects. To our knowledge, there is no reported clinical studies on the use of SCPC material to graft a pneumatized maxillary sinus. This aim of this current study is to compare SCPC to commonly used xenograft material in an augmented maxillary sinus.

DETAILED DESCRIPTION:
1. To assess the quality and quantity of the maxillary sinus bone prior to the placement of dental implants and subsequent restorations, approximately 20 patients will be randomly assigned to receive an augmentation of the maxillary sinus region using either Shefabone (synthetic bone) or Bio-Oss (xenograft).
2. With the use of pre-operative and post-operative limited view CBCT (cone-beam computed tomography) radiography, the maxillary sinus bone density will be assessed and compared between the individuals receiving Shefabone and the individuals receiving xenograft material.
3. Histomorphometric analysis will be used to assess, compare and contrast the quality and the quantity of the new vital bone cells generated when using these different graft materials.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 75 years of age
* at least one maxillary edentulous posterior site requiring maxillary sinus grafting and replacement with a dental implant.

Exclusion Criteria:

* current smokers/tobacco users
* are pregnant
* have active periodontal disease
* have uncontrolled diabetes
* have any autoimmune disease
* have kidney disease
* have liver disease
* are receiving radiation or chemotherapy
* have any type of radiographic periapical pathology such as a periapical abscess.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohanad Al-Sabbagh, DDS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Beneficial information for further research around the topic and/or information that may aid/benefit subjects or dentists in treatment may be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 participants were consented for the study but 2 did not meet eligibility criteria and did not receive an intervention
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 15 | 7
Completed | 14 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (12.4) | 63.4 (9.9) | 62.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 6 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Bone Density - Limited View CBCT (Cone-beam Computed Tomography) Measurements
Description: Bone density will be measured by limited view CBCT radiography pre- and post-operatively.
Time Frame: 5 months
Population: Data was incomplete for 4 subjects due to poor diagnostic quality or missed appointment
Measure: Mean (Standard Deviation); unit: percentage of bone height shrinkage
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 10 | 7
percentage of bone height shrinkage | 14.4 (3.9) | 1.5 (8.0)

2. Secondary Outcome: Bone Quality
Description: Bone quality will be measured using histomorphometric analysis.
Time Frame: 5.5 months
Population: Data was incomplete for 4 subjects due to poor diagnostic quality or missed appointment
Measure: Mean (Standard Deviation); unit: percentage of mineralized bone formation
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 10 | 7
percentage of mineralized bone formation | 60 (0) | 100 (0)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 0/14 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT04433117/Prot_SAP_001.pdf